CLINICAL TRIAL: NCT02515942
Title: A Randomized, Multi-Center, Single Masked, Sham Controlled, Proof-of-Concept Study of Intravitreal CLG561 as a Monotherapy and in Combination With LFG316 in Subjects With Geographic Atrophy
Brief Title: CLG561 Proof-of-Concept Study as a Monotherapy and in Combination With LFG316 in Subjects With Geographic Atrophy (GA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Novartis Institutes for BioMedical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLG561-2201; CCLG561X2201 (Other: Novartis Institutes for BioMedical Research)
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Geographic Atrophy
Keywords: Geographic atrophy (GA); Macular degeneration; Dry age-related macular degeneration (AMD); Intravitreal (IVT); Retinal diseases; Fundus auto fluorescence (FAF)
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration; Retinal Diseases | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CLG561 (Experimental): CLG561 10 mg, one IVT injection every 28 days for a total of 12 injections
  Interventions: Drug: CLG561
- CLG561+LFG316 (Experimental): CLG561 5mg + LFG316 5 mg, one IVT injection every 28 days for a total of 12 injections
  Interventions: Drug: CLG561; Drug: LFG316
- Sham Injection (Sham Comparator): One sham injection every 28 days for total of 12 sham injections
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: CLG561
  Arms: CLG561; CLG561+LFG316
Drug: LFG316
  Arms: CLG561+LFG316
Drug: Sham injection — Empty syringe (without a needle) placed against the eye
  Arms: Sham Injection

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 12 (every 28 days) intravitreal (IVT) injections of CLG561 as a monotherapy and in combination with LFG316 as compared to sham in subjects with geographic atrophy.

DETAILED DESCRIPTION:
This study consists of an up-to 30-day screening period, an approximately 336-day treatment period, and a follow-up period consisting of two visits occurring 4 and 16 weeks after the last administered injection.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent form;
* Geographic atrophy in both eyes;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Pregnant or lactating women and women of child-bearing potential;
* Any medical condition (systemic or ophthalmic) that may preclude the safe administration of test article or safe participation in this study;
* Any contraindications or hypersensitivities to any component of the LFG316 or CLG561 solution;
* Any contraindications to IVT injections;
* Ocular surgery in either eye within 90 days of screening;
* Uncontrolled ocular hypertension or glaucoma in the study eye;
* Other protocol-specified exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-09-25 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr Clinical Manager, Pharma, GCRA, Study Director — Alcon Research

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 28 sites in the US and Puerto Rico.
Pre-assignment Details: This reporting group includes all randomized participants.
Groups:
- CLG561: CLG561 10 mg, one intravitreal (IVT) injection every 28 days for a total of 12 injections
- CLG561+LFG316: CLG561 5 mg +LFG316 5 mg, one IVT injection every 28 days for a total of 12 injections
Period: Overall Study
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Started | 36 | 39 | 39
Safety Analysis Set (All subjects who received any study drug) | 36 | 39 | 39
Full Analysis Set (FAS) (Subjects who received study treatment & at least 1 follow-up visit with assessment of GA lesion size) | 35 | 37 | 38
Per Protocol Analysis Set (PPS) (FAS with no critical protocol deviations & with a valid assessment of primary efficacy endpoint) | 30 | 35 | 34
Pharmacokinetics (PK) Analysis Set (Subjects in safety set with evaluable PK data & no major protocol deviations that impacted PK data) | 36 | 39 | 0
Completed Day 85 | 35 | 38 | 37
Completed Day 169 | 32 | 37 | 37
Completed Day 253 | 29 (One subject missed Day 253 visit) | 37 | 36
Completed Day 337 | 30 | 36 | 35
Completed | 29 | 36 | 35
Not Completed | 7 | 3 | 4
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- CLG561+LFG316: CLG561 5 mg + LFG316 5 mg, one IVT injection every 28 days for a total of 12 injections
- Total: Total of all reporting groups
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection | Total
Number analyzed (Participants) | 36 | 39 | 39 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (8.61) | 78.8 (7.11) | 78.7 (9.80) | 78.4 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 24 | 67
  Male | 14 | 18 | 15 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 5 | 13
  Not Hispanic or Latino | 31 | 35 | 33 | 99
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 38 | 38
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 35 | 39 | 0 | 74
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Serious Adverse Event That, in the Opinion of the Investigator, is Related to the Study Drug
Description: A serious adverse event (SAE) was defined as any adverse experience that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event. All SAEs related to the study drug are reported. No statistical analysis was conducted.
Time Frame: Up to Day 421
Population: Safety Analysis Set
Measure: Number; unit: subjects
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 36 | 39 | 39
subjects | 0 | 0 | 0

2. Primary Outcome: Mean Change From Baseline in Intraocular Pressure (IOP)
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry and reported in millimeters of mercury (mmHg). A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). Baseline is defined as the last measurement prior to first dose of treatment. A more negative change indicates a greater amount of improvement. One eye (study eye) contributed to the analysis. No statistical analysis was conducted.
Time Frame: Baseline (Day 1), Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225, Day 253, Day 281, Day 309
Population: Safety Analysis Set. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 36 | 39 | 39
mmHg
  Baseline (BL) (Day 1) | 15.1 (3.58) | 14.5 (3.42) | 15.5 (3.54)
  Change from BL at Day 29: number analyzed (Participants) | 35 | 39 | 39
  Change from BL at Day 29 | -0.2 (2.57) | 0.0 (2.95) | -0.7 (3.74)
  Change from BL at Day 57: number analyzed (Participants) | 36 | 39 | 38
  Change from BL at Day 57 | -0.2 (3.46) | -0.4 (2.70) | -0.1 (3.06)
  Change from BL at Day 85: number analyzed (Participants) | 35 | 38 | 37
  Change from BL at Day 85 | -0.1 (2.80) | -0.1 (3.02) | 0.2 (2.86)
  Change from BL at Day 113: number analyzed (Participants) | 35 | 37 | 38
  Change from BL at Day 113 | 0.2 (3.84) | 0.4 (3.31) | -0.7 (2.69)
  Change from BL at Day 141: number analyzed (Participants) | 32 | 38 | 37
  Change from BL at Day 141 | 0.4 (2.93) | 0.1 (3.82) | -0.6 (3.09)
  Change from BL at Day 169: number analyzed (Participants) | 32 | 37 | 37
  Change from BL at Day 169 | 0.4 (4.35) | -0.1 (3.33) | -0.6 (3.75)
  Change from BL at Day 197: number analyzed (Participants) | 33 | 37 | 37
  Change from BL at Day 197 | -0.4 (3.88) | -0.0 (3.74) | -0.2 (3.13)
  Change from BL at Day 225: number analyzed (Participants) | 32 | 36 | 37
  Change from BL at Day 225 | -0.3 (3.72) | -0.0 (4.11) | -0.4 (3.40)
  Change from BL at Day 253: number analyzed (Participants) | 29 | 37 | 36
  Change from BL at Day 253 | 0.6 (4.39) | -0.2 (3.61) | -1.1 (3.75)
  Change from BL at Day 281: number analyzed (Participants) | 30 | 37 | 34
  Change from BL at Day 281 | 1.6 (8.32) | 0.5 (3.72) | -0.6 (3.91)
  Change from BL at Day 309: number analyzed (Participants) | 30 | 36 | 35
  Change from BL at Day 309 | 1.0 (2.97) | 0.0 (3.43) | -1.2 (4.00)

3. Primary Outcome: Change in GA Lesion Size From Baseline to Day 337 as Measured by Fundus Autofluorescence (FAF)
Description: Geographic atrophy, also known as atrophic age-related macular degeneration (AMD) or advanced dry AMD, is an advanced form of age-related macular degeneration that can result in the progressive and irreversible loss of retina which can lead to a loss of visual function over time. Geographic atrophy (GA) lesion size was assessed by a Central Reading Center (CRC) using FAF. Baseline is defined as the last measurement prior to first dose of treatment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 1), Day 337
Population: PPS. Only subjects with a value at both baseline and that time point are included.
Measure: Least Squares Mean (80% Confidence Interval); unit: square millimeters (mm2)
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 29 | 34 | 33
square millimeters (mm2) | 1.53 [1.31 to 1.74] | 1.88 [1.68 to 2.08] | 1.82 [1.61 to 2.03]
Statistical Analysis 1: Comparison: CLG561 vs CLG561+LFG316; Test type: Superiority — Least squares mean for change from baseline from ANCOVA model with treatment, baseline lesion location (foveal vs. extrafoveal), baseline lesion type (unifocal vs. multifocal), baseline lesion size as covariates after multiple imputations; p = 0.0636, ANCOVA; Treatment Effect = -0.35, 80% CI 2-sided [-0.64 to -0.06]
Statistical Analysis 2: Comparison: CLG561 vs Sham Injection; Least squares mean for change from baseline from ANCOVA model with treatment, baseline lesion location (foveal vs. extrafoveal), baseline lesion type (unifocal vs. multifocal), baseline lesion size as covariates after multiple imputations; Test type: Superiority; p = 0.1019, ANCOVA; Treatment Effect = -0.29, 80% CI 2-sided [-0.59 to 0.00]
Statistical Analysis 3: Comparison: CLG561+LFG316 vs Sham Injection; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.5987, ANCOVA; Treatment Effect = 0.06, 80% CI 2-sided [-0.24 to 0.35]

4. Secondary Outcome: Change in GA Lesion Size From Baseline to Day 85, 169, and 253 as Measured by FAF
Description: as for outcome 3
Time Frame: Baseline (Day 1), Day 85, Day 169, Day 253
Population: PPS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Least Squares Mean (80% Confidence Interval); unit: mm2
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 30 | 35 | 34
mm2
  Change from BL at Day 85: number analyzed (Participants) | 28 | 32 | 32
  Change from BL at Day 85 | 0.41 [0.33 to 0.49] | 0.41 [0.34 to 0.48] | 0.37 [0.30 to 0.45]
  Change from BL at Day 169: number analyzed (Participants) | 29 | 33 | 32
  Change from BL at Day 169 | 0.69 [0.58 to 0.80] | 0.81 [0.71 to 0.92] | 0.82 [0.72 to 0.93]
  Change from BL at Day 253: number analyzed (Participants) | 28 | 34 | 33
  Change from BL at Day 253 | 1.08 [0.93 to 1.22] | 1.33 [1.20 to 1.46] | 1.25 [1.11 to 1.38]
Statistical Analysis 1: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 85; Test type: Superiority — Least squares mean for change from baseline from repeated measures mixed effect model with treatment, visit and treatment*visit interaction, baseline lesion location (foveal vs. extrafoveal), baseline lesion type (unifocal vs. multifocal) and baseline value as fixed effects, and unstructured covariance for observations within the same subject; p = 0.5029, Mixed Models Analysis; Treatment Effect = 0.00, 80% CI 2-sided [-0.11 to 0.11]
Statistical Analysis 2: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6820, Mixed Models Analysis; Treatment Effect = 0.04, 80% CI 2-sided [-0.07 to 0.14]
Statistical Analysis 3: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6826, Mixed Models Analysis; Treatment Effect = 0.04, 80% CI 2-sided [-0.07 to 0.14]
Statistical Analysis 4: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1545, Mixed Models Analysis; Treatment Effect = -0.12, 80% CI 2-sided [-0.28 to 0.03]
Statistical Analysis 5: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1398, Mixed Models Analysis; Treatment Effect = -0.13, 80% CI 2-sided [-0.29 to 0.02]
Statistical Analysis 6: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4717, Mixed Models Analysis; Treatment Effect = -0.01, 80% CI 2-sided [-0.16 to 0.14]
Statistical Analysis 7: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0530, Mixed Models Analysis; Treatment Effect = -0.25, 80% CI 2-sided [-0.45 to -0.05]
Statistical Analysis 8: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1386, Mixed Models Analysis; Treatment Effect = -0.17, 80% CI 2-sided [-0.37 to 0.03]
Statistical Analysis 9: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7087, Mixed Models Analysis; Treatment Effect = 0.08, 80% CI 2-sided [-0.11 to 0.27]

5. Secondary Outcome: Mean Change in GA Lesion Size From Baseline to Day 421 as Measured by FAF
Description: Geographic atrophy, also known as atrophic age-related macular degeneration (AMD) or advanced dry AMD, is an advanced form of age-related macular degeneration that can result in the progressive and irreversible loss of retina which can lead to a loss of visual function over time. Geographic atrophy (GA) lesion size was assessed by a Central Reading Center (CRC) using FAF. Baseline is defined as the last measurement prior to first dose of treatment. One eye (study eye) contributed to the analysis. Day 421 measurements were only summarized descriptively and did not include any statistical modeling.
Time Frame: Baseline (Day 1), Day 421
Population: PPS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 30 | 35 | 34
mm2
  Baseline (Day 1) | 9.090 (3.9628) | 9.070 (3.6955) | 9.017 (4.2132)
  Change from Baseline at Day 421: number analyzed (Participants) | 28 | 32 | 31
  Change from Baseline at Day 421 | 2.056 (1.0618) | 2.449 (1.0691) | 2.395 (1.1905)

6. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline by Visit up to Day 337 as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS)
Description: BCVA was assessed using ETDRS testing at 4 meters. Baseline is defined as the last measurement prior to first dose of treatment. BCVA change was defined as a change in letters read from the baseline assessment. A positive change value indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 1), Day 2, Day 8, Day 15, Day 29, Day 30, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225, Day 253, Day 281, Day 309, Day 337
Population: FAS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Least Squares Mean (80% Confidence Interval); unit: letters
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 35 | 37 | 38
letters
  Change from BL at Day 2: number analyzed (Participants) | 34 | 35 | 36
  Change from BL at Day 2 | -0.93 [-2.65 to 0.78] | 1.79 [0.09 to 3.48] | -1.44 [-3.10 to 0.22]
  Change from BL at Day 8: number analyzed (Participants) | 33 | 35 | 37
  Change from BL at Day 8 | 2.14 [0.31 to 3.98] | 2.46 [0.67 to 4.26] | 0.86 [-0.88 to 2.60]
  Change from BL at Day 15: number analyzed (Participants) | 32 | 35 | 37
  Change from BL at Day 15 | 2.89 [1.10 to 4.69] | 4.83 [3.10 to 6.55] | 3.02 [1.33 to 4.70]
  Change from BL at Day 29: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 29 | 3.28 [1.53 to 5.02] | 5.29 [3.61 to 6.96] | 1.25 [-0.40 to 2.90]
  Change from BL at Day 30: number analyzed (Participants) | 32 | 35 | 36
  Change from BL at Day 30 | 3.30 [1.70 to 4.91] | 3.16 [1.62 to 4.71] | 2.92 [1.40 to 4.44]
  Change from BL at Day 57: number analyzed (Participants) | 34 | 36 | 36
  Change from BL at Day 57 | 3.65 [1.74 to 5.55] | 4.69 [2.84 to 6.54] | 4.25 [2.42 to 6.08]
  Change from BL at Day 85: number analyzed (Participants) | 34 | 35 | 36
  Change from BL at Day 85 | 3.86 [2.05 to 5.68] | 2.57 [0.80 to 4.35] | 3.05 [1.31 to 4.80]
  Change from BL at Day 113: number analyzed (Participants) | 34 | 34 | 37
  Change from BL at Day 113 | 3.09 [1.11 to 5.07] | 3.60 [1.65 to 5.54] | 3.40 [1.50 to 5.29]
  Change from BL at Day 141: number analyzed (Participants) | 33 | 35 | 37
  Change from BL at Day 141 | 3.20 [1.28 to 5.12] | 5.14 [3.27 to 7.01] | 2.22 [0.39 to 4.05]
  Change from BL at Day 169: number analyzed (Participants) | 31 | 36 | 36
  Change from BL at Day 169 | 2.62 [0.64 to 4.60] | 3.57 [1.67 to 5.47] | 3.61 [1.73 to 5.48]
  Change from BL at Day 197: number analyzed (Participants) | 32 | 35 | 36
  Change from BL at Day 197 | 2.30 [0.05 to 4.54] | 2.60 [0.42 to 4.77] | 3.54 [1.41 to 5.67]
  Change from BL at Day 225: number analyzed (Participants) | 31 | 34 | 36
  Change from BL at Day 225 | 2.98 [0.54 to 5.41] | 3.33 [0.98 to 5.68] | 1.87 [-0.43 to 4.17]
  Change from BL at Day 253: number analyzed (Participants) | 28 | 35 | 35
  Change from BL at Day 253 | 2.76 [0.18 to 5.34] | 3.31 [0.85 to 5.77] | 0.46 [-1.96 to 2.88]
  Change from BL at Day 281: number analyzed (Participants) | 29 | 35 | 34
  Change from BL at Day 281 | 1.52 [-1.17 to 4.21] | 2.08 [-0.48 to 4.63] | 0.67 [-1.86 to 3.20]
  Change from BL at Day 309: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Day 309 | 1.39 [-1.24 to 4.01] | 2.92 [0.43 to 5.42] | -0.75 [-3.22 to 1.71]
  Change from BL at Day 337: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Day 337 | 0.25 [-2.92 to 3.42] | 0.07 [-2.93 to 3.08] | 0.45 [-2.52 to 3.41]
Statistical Analysis 1: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.9243, Mixed Models Analysis; Treatment Effect = -2.72, 80% CI 2-sided [-5.15 to -0.29]
Statistical Analysis 2: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3929, Mixed Models Analysis; Treatment Effect = 0.51, 80% CI 2-sided [-1.89 to 2.91]
Statistical Analysis 3: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0418, Mixed Models Analysis; Treatment Effect = 3.23, 80% CI 2-sided [0.85 to 5.61]
Statistical Analysis 4: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 8; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5632, Mixed Models Analysis; Treatment Effect = -0.32, 80% CI 2-sided [-2.91 to 2.27]
Statistical Analysis 5: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 8; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2575, Mixed Models Analysis; Treatment Effect = 1.29, 80% CI 2-sided [-1.25 to 3.83]
Statistical Analysis 6: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 8; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2058, Mixed Models Analysis; Treatment Effect = 1.61, 80% CI 2-sided [-0.91 to 4.12]
Statistical Analysis 7: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 15; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.8392, Mixed Models Analysis; Treatment Effect = -1.94, 80% CI 2-sided [-4.44 to 0.57]
Statistical Analysis 8: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 15; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5255, Mixed Models Analysis; Treatment Effecgt = -0.12, 80% CI 2-sided [-2.59 to 2.35]
Statistical Analysis 9: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 15; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1685, Mixed Models Analysis; Treatment Effect = 1.81, 80% CI 2-sided [-0.61 to 4.24]
Statistical Analysis 10: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.8544, Mixed Models Analysis; Treatment = -2.01, 80% CI 2-sided [-4.45 to 0.43]
Statistical Analysis 11: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1402, Mixed Models Analysis; Treatment Effect = 2.03, 80% CI 2-sided [-0.38 to 4.44]
Statistical Analysis 12: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0150, Mixed Models Analysis; Treatment Effect = 4.03, 80% CI 2-sided [1.67 to 6.40]
Statistical Analysis 13: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 30; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4682, Mixed Models Analysis; Treatment Effect = 0.14, 80% CI 2-sided [-2.11 to 2.39]
Statistical Analysis 14: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 30; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4125, Mixed Models Analysis; Treatment Effect = 0.38, 80% CI 2-sided [-1.84 to 2.60]
Statistical Analysis 15: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 30; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4431, Mixed Models Analysis; Treatment Effect = 0.24, 80% CI 2-sided [-1.94 to 2.42]
Statistical Analysis 16: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6924, Mixed Models Analysis; Treatment Effect = -1.04, 80% CI 2-sided [-3.72 to 1.63]
Statistical Analysis 17: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6160, Mixed Models Analysis; Treatment Effect = -0.61, 80% CI 2-sided [-3.26 to 2.04]
Statistical Analysis 18: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4149, Mixed Models Analysis; Treatment Effect = 0.44, 80% CI 2-sided [-2.18 to 3.06]
Statistical Analysis 19: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2582, Mixed Models Analysis; Treatment Effect = 1.29, 80% CI 2-sided [-1.27 to 3.85]
Statistical Analysis 20: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3402, Mixed Models Analysis; Treatment Effect = 0.81, 80% CI 2-sided [-1.72 to 3.34]
Statistical Analysis 21: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5976, Mixed Models Analysis; Treatment Effect = -0.48, 80% CI 2-sided [-2.99 to 2.03]
Statistical Analysis 22: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5916, Mixed Models Analysis; Treatment Effect = -0.50, 80% CI 2-sided [-3.30 to 2.29]
Statistical Analysis 23: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5564, Mixed Models Analysis; Treatment Effect = -0.30, 80% CI 2-sided [-3.05 to 2.45]
Statistical Analysis 24: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4625, Mixed Models Analysis; Treatment Effect = 0.20, 80% CI 2-sided [-2.53 to 2.93]
Statistical Analysis 25: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.8221, Mixed Models Analysis; Treatment Effect = -1.94, 80% CI 2-sided [-4.64 to 0.76]
Statistical Analysis 26: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3179, Mixed Models Analysis; Treatment Effect = 0.98, 80% CI 2-sided [-1.68 to 3.64]
Statistical Analysis 27: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0773, Mixed Models Analysis; Treatment Effect = 2.92, 80% CI 2-sided [0.29 to 5.55]
Statistical Analysis 28: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6708, Mixed Models Analysis; Treatment Effect = -0.95, 80% CI 2-sided [-3.71 to 1.81]
Statistical Analysis 29: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6790, Mixed Models Analysis; Treatment Effect = -0.99, 80% CI 2-sided [-3.71 to 1.74]
Statistical Analysis 30: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5070, Mixed Models Analysis; Treatment Effect = -0.04, 80% CI 2-sided [-2.72 to 2.64]
Statistical Analysis 31: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5487, Mixed Models Analysis; Treatment Effect = -0.30, 80% CI 2-sided [-3.44 to 2.84]
Statistical Analysis 32: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6973, Mixed Models Analysis; Treatment Effect = -1.25, 80% CI 2-sided [-4.35 to 1.85]
Statistical Analysis 33: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6548, Mixed Models Analysis; Treatment Effect = -0.95, 80% CI 2-sided [-4.00 to 2.11]
Statistical Analysis 34: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5533, Mixed Models Analysis; Treatment Effect = -0.35, 80% CI 2-sided [-3.76 to 3.05]
Statistical Analysis 35: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3358, Mixed Models Analysis; Treatment Effect = 1.11, 80% CI 2-sided [-2.25 to 4.46]
Statistical Analysis 36: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2850, Mixed Models Analysis; Treatment Effect = 1.46, 80% CI 2-sided [-1.85 to 4.77]
Statistical Analysis 37: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5778, Mixed Models Analysis; Treatment Effect = -0.55, 80% CI 2-sided [-4.14 to 3.04]
Statistical Analysis 38: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2018, Mixed Models Analysis; Treatment Effect = 2.30, 80% CI 2-sided [-1.24 to 5.85]
Statistical Analysis 39: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1457, Mixed Models Analysis; Treatment Effect = 2.85, 80% CI 2-sided [-0.62 to 6.32]
Statistical Analysis 40: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5758, Mixed Models Analysis; Treatment Effect = -0.56, 80% CI 2-sided [-4.29 to 3.18]
Statistical Analysis 41: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3833, Mixed Models Analysis; Treatment Effect = 0.85, 80% CI 2-sided [-2.84 to 4.55]
Statistical Analysis 42: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3083, Mixed Models Analysis; Treatment Effect = 1.41, 80% CI 2-sided [-2.21 to 5.02]
Statistical Analysis 43: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7063, Mixed Models Analysis; Treatment Effect = -1.54, 80% CI 2-sided [-5.19 to 2.11]
Statistical Analysis 44: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2227, Mixed Models Analysis; Treatment Effect = 2.14, 80% CI 2-sided [-1.46 to 5.74]
Statistical Analysis 45: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0907, Mixed Models Analysis; Treatment Effect = 3.68, 80% CI 2-sided [0.15 to 7.21]
Statistical Analysis 46: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4799, Mixed Models Analysis; Treatment Effect = 0.17, 80% CI 2-sided [-4.23 to 4.57]
Statistical Analysis 47: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5237, Mixed Models Analysis; Treatment Effect = -0.20, 80% CI 2-sided [-4.54 to 4.14]
Statistical Analysis 48: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5451, Mixed Models Analysis; Treatment Effect = -0.37, 80% CI 2-sided [-4.62 to 3.87]

7. Secondary Outcome: Change in Low Luminance Visual Acuity (LLVA) From Baseline up to Day 337 as Measured by ETDRS
Description: Low Luminance Visual Acuity (VA) was assessed using ETDRS testing at 4 meters with a neutral density filter to reduce chart luminance to 3 candelas/m2. Baseline is defined as the last measurement prior to first dose of treatment. BCVA change was defined as a change in letters read from the baseline assessment. A positive change value indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 1), Day 2, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 225, Day 253, Day 281, Day 309, Day 337
Population: FAS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Least Squares Mean (80% Confidence Interval); unit: letters
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 35 | 37 | 38
letters
  Change from BL at Day 2: number analyzed (Participants) | 34 | 34 | 36
  Change from BL at Day 2 | -0.57 [-1.93 to 0.79] | -0.72 [-2.09 to 0.65] | -1.03 [-2.36 to 0.29]
  Change from BL at Day 29: number analyzed (Participants) | 33 | 35 | 36
  Change from BL at Day 29 | 0.99 [-0.71 to 2.69] | 3.87 [2.21 to 5.53] | 1.39 [-0.23 to 3.02]
  Change from BL at Day 57: number analyzed (Participants) | 34 | 35 | 36
  Change from BL at Day 57 | 2.41 [0.40 to 4.43] | 1.89 [-0.11 to 3.88] | 1.18 [-0.78 to 3.13]
  Change from BL at Day 85: number analyzed (Participants) | 34 | 34 | 36
  Change from BL at Day 85 | 3.80 [1.86 to 5.75] | 2.89 [0.96 to 4.83] | -0.15 [-2.03 to 1.73]
  Change from BL at Day 113: number analyzed (Participants) | 34 | 33 | 37
  Change from BL at Day 113 | 3.59 [1.52 to 5.65] | -0.09 [-2.16 to 1.98] | 1.67 [-0.31 to 3.65]
  Change from BL at Day 141: number analyzed (Participants) | 32 | 33 | 37
  Change from BL at Day 141 | 2.90 [0.36 to 5.44] | 1.41 [-1.10 to 3.93] | 1.57 [-0.85 to 3.99]
  Change from BL at Day 169: number analyzed (Participants) | 31 | 35 | 36
  Change from BL at Day 169 | 1.40 [-0.68 to 3.47] | 3.03 [1.01 to 5.05] | 2.78 [0.81 to 4.75]
  Change from BL at Day 197: number analyzed (Participants) | 32 | 34 | 36
  Change from BL at Day 197 | 2.52 [0.20 to 4.83] | 2.23 [-0.05 to 4.50] | 1.58 [-0.62 to 3.78]
  Change from BL at Day 225: number analyzed (Participants) | 31 | 33 | 36
  Change from BL at Day 225 | 2.47 [-0.20 to 5.14] | 0.69 [-1.94 to 3.32] | 0.75 [-1.79 to 3.29]
  Change from BL at Day 253: number analyzed (Participants) | 28 | 34 | 35
  Change from BL at Day 253 | 3.50 [0.95 to 6.04] | 0.68 [-1.76 to 3.12] | 1.71 [-0.67 to 4.08]
  Change from BL at Day 281: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Day 281 | 3.21 [0.30 to 6.12] | 1.90 [-0.93 to 4.73] | 0.79 [-1.96 to 3.55]
  Change from BL at Day 309: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Day 309 | 1.72 [-1.12 to 4.56] | 1.79 [-0.96 to 4.53] | -0.61 [-3.29 to 2.06]
  Change from BL at Day 337: number analyzed (Participants) | 29 | 33 | 34
  Change from BL at Day 337 | 1.47 [-1.38 to 4.32] | -1.09 [-3.85 to 1.68] | -0.73 [-3.42 to 1.96]
Statistical Analysis 1: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4609, Mixed Models Analysis; Treatment Effect = 0.15, 80% CI 2-sided [-1.79 to 2.09]
Statistical Analysis 2: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3771, Mixed Models Analysis; Treatment Effect = 0.46, 80% CI 2-sided [-1.44 to 2.37]
Statistical Analysis 3: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4161, Mixed Models Analysis; Treatment Effect = 0.32, 80% CI 2-sided [-1.60 to 2.24]
Statistical Analysis 4: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.9385, Mixed Models Analysis; Treatment Effect = -2.88, 80% CI 2-sided [-5.26 to -0.49]
Statistical Analysis 5: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5862, Mixed Models Analysis; Treatment Effect = -0.40, 80% CI 2-sided [-2.76 to 1.96]
Statistical Analysis 6: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0875, Mixed Models Analysis; Treatment Effect = 2.48, 80% CI 2-sided [0.14 to 4.82]
Statistical Analysis 7: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4059, Mixed Models Analysis; Treatment Effect = 0.53, 80% CI 2-sided [-2.32 to 3.37]
Statistical Analysis 8: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2860, Mixed Models Analysis; Treatment Effect = 1.24, 80% CI 2-sided [-1.58 to 4.05]
Statistical Analysis 9: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3727, Mixed Models Analysis; Treatment Effect = 0.71, 80% CI 2-sided [-2.10 to 3.52]
Statistical Analysis 10: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3360, Mixed Models Analysis; Treatment Effect = 0.91, 80% CI 2-sided [-1.85 to 3.66]
Statistical Analysis 11: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0316, Mixed Models Analysis; Treatment Effect = 3.95, 80% CI 2-sided [1.24 to 6.66]
Statistical Analysis 12: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0762, Mixed Models Analysis; Treatment Effect = 3.04, 80% CI 2-sided [0.32 to 5.76]
Statistical Analysis 13: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0544, Mixed Models Analysis; Treatment Effect = 3.68, 80% CI 2-sided [0.75 to 6.61]
Statistical Analysis 14: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1955, Mixed Models Analysis; Treatment Effect = 1.91, 80% CI 2-sided [-0.95 to 4.77]
Statistical Analysis 15: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7844, Mixed Models Analysis; Treatment Effect = -1.77, 80% CI 2-sided [-4.65 to 1.12]
Statistical Analysis 16: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2973, Mixed Models Analysis; Treatment Effect = 1.49, 80% CI 2-sided [-2.11 to 5.08]
Statistical Analysis 17: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3127, Mixed Models Analysis; Treatment Effect = 1.33, 80% CI 2-sided [-2.18 to 4.84]
Statistical Analysis 18: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5227, Mixed Models Analysis; Treatment Effect = -0.16, 80% CI 2-sided [-3.67 to 3.36]
Statistical Analysis 19: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7643, Mixed Models Analysis; Treatment Effect = -1.63, 80% CI 2-sided [-4.54 to 1.28]
Statistical Analysis 20: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7331, Mixed Models Analysis; Treatment Effect = -1.38, 80% CI 2-sided [-4.25 to 1.48]
Statistical Analysis 21: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4557, Mixed Models Analysis; Treatment Effect = 0.25, 80% CI 2-sided [-2.59 to 3.09]
Statistical Analysis 22: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4549, Mixed Models Analysis; Treatment Effect = 0.29, 80% CI 2-sided [-2.97 to 3.55]
Statistical Analysis 23: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3535, Mixed Models Analysis; Treatment Effect = 0.93, 80% CI 2-sided [-2.26 to 4.13]
Statistical Analysis 24: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3970, Mixed Models Analysis; Treatment Effect = 0.65, 80% CI 2-sided [-2.54 to 3.84]
Statistical Analysis 25: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2714, Mixed Models Analysis; Treatment Effect = 1.78, 80% CI 2-sided [-1.99 to 5.55]
Statistical Analysis 26: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2741, Mixed Models Analysis; Treatment Effect = 1.72, 80% CI 2-sided [-1.97 to 5.41]
Statistical Analysis 27: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5084, Mixed Models Analysis; Treatment Effect = -0.06, 80% CI 2-sided [-3.74 to 3.62]
Statistical Analysis 28: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1537, Mixed Models Analysis; Treatment Effect = 2.82, 80% CI 2-sided [-0.73 to 6.37]
Statistical Analysis 29: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2542, Mixed Models Analysis; Treatment Effect = 1.79, 80% CI 2-sided [-1.69 to 5.27]
Statistical Analysis 30: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6504, Mixed Models Analysis; Treatment Effect = -1.03, 80% CI 2-sided [-4.46 to 2.40]
Statistical Analysis 31: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3405, Mixed Models Analysis; Treatment Effect = 1.30, 80% CI 2-sided [-2.78 to 5.38]
Statistical Analysis 32: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2194, Mixed Models Analysis; Treatment Effect = 2.41, 80% CI 2-sided [-1.59 to 6.42]
Statistical Analysis 33: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3596, Mixed Models Analysis; Treatment Effect = 1.11, 80% CI 2-sided [-2.87 to 5.09]
Statistical Analysis 34: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5086, Mixed Models Analysis; Treatment Effect = -0.07, 80% CI 2-sided [-4.04 to 3.90]
Statistical Analysis 35: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2211, Mixed Models Analysis; Treatment Effect = 2.33, 80% CI 2-sided [-1.57 to 6.23]
Statistical Analysis 36: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2126, Mixed Models Analysis; Treatment Effect = 2.40, 80% CI 2-sided [-1.47 to 6.26]
Statistical Analysis 37: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2053, Mixed Models Analysis; Treatment Effect = 2.56, 80% CI 2-sided [-1.44 to 6.55]
Statistical Analysis 38: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2353, Mixed Models Analysis; Treatment Effect = 2.20, 80% CI 2-sided [-1.72 to 6.12]
Statistical Analysis 39: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5471, Mixed Models Analysis; Treatment Effect = -0.36, 80% CI 2-sided [-4.24 to 3.53]

8. Secondary Outcome: Change in LLVA Deficit From Baseline up to Day 337 as Measured by ETDRS
Description: Low Luminance Visual Acuity (VA) was assessed using ETDRS testing at 4 meters with a neutral density filter to reduce chart luminance to 3 candelas/m2. A deficit in LLVA is defined as a loss in letters read from baseline. Baseline is defined as the last measurement prior to first dose of treatment. A negative change value indicates improvement (more letters read). One eye (study eye) contributed to the analysis.
Time Frame: as for outcome 7
Population: FAS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Least Squares Mean (80% Confidence Interval); unit: letters
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 35 | 37 | 38
letters
  Change from BL at Day 2: number analyzed (Participants) | 34 | 34 | 36
  Change from BL at Day 2 | -0.43 [-2.28 to 1.43] | 2.32 [0.45 to 4.18] | -0.15 [-1.96 to 1.67]
  Change from BL at Day 29: number analyzed (Participants) | 33 | 35 | 36
  Change from BL at Day 29 | 2.43 [0.54 to 4.32] | 1.27 [-0.57 to 3.12] | 0.06 [-1.76 to 1.88]
  Change from BL at Day 57: number analyzed (Participants) | 34 | 35 | 36
  Change from BL at Day 57 | 1.38 [-0.79 to 3.55] | 2.54 [0.40 to 4.69] | 3.07 [0.97 to 5.18]
  Change from BL at Day 85: number analyzed (Participants) | 34 | 34 | 36
  Change from BL at Day 85 | -0.10 [-2.01 to 1.81] | -0.23 [-2.14 to 1.68] | 3.27 [1.41 to 5.13]
  Change from BL at Day 113: number analyzed (Participants) | 34 | 33 | 37
  Change from BL at Day 113 | -0.33 [-2.58 to 1.92] | 3.59 [1.34 to 5.85] | 1.83 [-0.34 to 3.99]
  Change from BL at Day 141: number analyzed (Participants) | 32 | 33 | 37
  Change from BL at Day 141 | 0.45 [-2.08 to 2.99] | 4.30 [1.79 to 6.81] | 0.83 [-1.58 to 3.25]
  Change from BL at Day 169: number analyzed (Participants) | 31 | 35 | 36
  Change from BL at Day 169 | 0.80 [-1.25 to 2.86] | 0.85 [-1.15 to 2.85] | 0.85 [-1.10 to 2.81]
  Change from BL at Day 197: number analyzed (Participants) | 32 | 34 | 36
  Change from BL at Day 197 | -0.37 [-2.62 to 1.88] | 0.72 [-1.49 to 2.93] | 2.08 [-0.07 to 4.23]
  Change from BL at Day 225: number analyzed (Participants) | 31 | 33 | 36
  Change from BL at Day 225 | -0.08 [-2.63 to 2.47] | 3.86 [1.35 to 6.36] | 1.39 [-1.04 to 3.82]
  Change from BL at Day 253: number analyzed (Participants) | 28 | 34 | 35
  Change from BL at Day 253 | -0.39 [-2.68 to 1.89] | 3.24 [1.06 to 5.42] | -0.85 [-2.99 to 1.28]
  Change from BL at Day 281: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Day 281 | -2.13 [-4.75 to 0.49] | 1.09 [-1.43 to 3.60] | 0.14 [-2.33 to 2.61]
  Change from BL at Day 309: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Day 309 | -0.62 [-3.26 to 2.01] | 2.02 [-0.53 to 4.56] | 0.07 [-2.42 to 2.57]
  Change from BL at Day 337: number analyzed (Participants) | 29 | 33 | 34
  Change from BL at Day 337 | -1.35 [-4.32 to 1.62] | 2.55 [-0.32 to 5.41] | 1.37 [-1.43 to 4.16]
Statistical Analysis 1: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0913, Mixed Models Analysis; Treatment Effect = -2.74, 80% CI 2-sided [-5.38 to -0.11]
Statistical Analysis 2: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4454, Mixed Models Analysis; Treatment Effect = -0.28, 80% CI 2-sided [-2.89 to 2.33]
Statistical Analysis 3: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 2; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.8861, Mixed Models Analysis; Treatment Effect = 2.46, 80% CI 2-sided [-0.16 to 5.08]
Statistical Analysis 4: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7130, Mixed Models Analysis; Treatment Effect = 1.16, 80% CI 2-sided [-1.49 to 3.80]
Statistical Analysis 5: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.8759, Mixed Models Analysis; Treatment Effect = 2.37, 80% CI 2-sided [-0.26 to 5.01]
Statistical Analysis 6: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 29; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7256, Mixed Models Analysis; Treatment Effect = 1.22, 80% CI 2-sided [-1.39 to 3.82]
Statistical Analysis 7: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3111, Mixed Models Analysis; Treatment Effect = -1.17, 80% CI 2-sided [-4.22 to 1.88]
Statistical Analysis 8: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2360, Mixed Models Analysis; Treatment Effect = -1.70, 80% CI 2-sided [-4.73 to 1.34]
Statistical Analysis 9: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 57; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4110, Mixed Models Analysis; Treatment Effect = -0.53, 80% CI 2-sided [-3.55 to 2.49]
Statistical Analysis 10: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5247, Mixed Models Analysis; Treatment Effect = 0.13, 80% CI 2-sided [-2.57 to 2.83]
Statistical Analysis 11: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0534, Mixed Models Analysis; Treatment Effect = -3.37, 80% CI 2-sided [-6.04 to -0.70]
Statistical Analysis 12: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 85; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0475, Mixed Models Analysis; Treatment Effect = -3.50, 80% CI 2-sided [-6.18 to -0.82]
Statistical Analysis 13: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0575, Mixed Models Analysis; Treatment Effect = -3.92, 80% CI 2-sided [-7.11 to -0.74]
Statistical Analysis 14: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1876, Mixed Models Analysis; Treatment Effect = -2.16, 80% CI 2-sided [-5.29 to 0.97]
Statistical Analysis 15: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 113; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7644, Mixed Models Analysis; Treatment Effect = 1.76, 80% CI 2-sided [-1.38 to 4.91]
Statistical Analysis 16: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0838, Mixed Models Analysis; Treatment Effect = -3.85, 80% CI 2-sided [-7.42 to -0.28]
Statistical Analysis 17: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4444, Mixed Models Analysis; Treatment Effect = -0.38, 80% CI 2-sided [-3.89 to 3.13]
Statistical Analysis 18: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 141; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.8977, Mixed Models Analysis; Treatment Effect = 3.47, 80% CI 2-sided [-0.04 to 6.97]
Statistical Analysis 19: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4917, Mixed Models Analysis; Treatment Effect = -0.05, 80% CI 2-sided [-2.92 to 2.82]
Statistical Analysis 20: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4909, Mixed Models Analysis; Treatment Effect = -0.05, 80% CI 2-sided [-2.89 to 2.79]
Statistical Analysis 21: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 169; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4992, Mixed Models Analysis; Treatment Effect = -0.00, 80% CI 2-sided [-2.82 to 2.81]
Statistical Analysis 22: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.3285, Mixed Models Analysis; Treatment Effect = -1.09, 80% CI 2-sided [-4.25 to 2.07]
Statistical Analysis 23: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1568, Mixed Models Analysis; Treatment Effect = -2.45, 80% CI 2-sided [-5.57 to 0.67]
Statistical Analysis 24: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 197; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2867, Mixed Models Analysis; Treatment Effect = -1.36, 80% CI 2-sided [-4.46 to 1.74]
Statistical Analysis 25: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0798, Mixed Models Analysis; Treatment Effect = -3.93, 80% CI 2-sided [-7.51 to -0.35]
Statistical Analysis 26: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2962, Mixed Models Analysis; Treatment Effect = -1.47, 80% CI 2-sided [-5.00 to 2.06]
Statistical Analysis 27: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 225; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.8163, Mixed Models Analysis; Treatment Effect = 2.46, 80% CI 2-sided [-1.05 to 5.98]
Statistical Analysis 28: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0708, Mixed Models Analysis; Treatment Effect = -3.64, 80% CI 2-sided [-6.81 to -0.47]
Statistical Analysis 29: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.5750, Mixed Models Analysis; Treatment Effect = 0.46, 80% CI 2-sided [-2.67 to 3.59]
Statistical Analysis 30: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 253; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.9560, Mixed Models Analysis; Treatment Effect = 4.10, 80% CI 2-sided [1.03 to 7.17]
Statistical Analysis 31: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1283, Mixed Models Analysis; Treatment Effect = -3.22, 80% CI 2-sided [-6.86 to 0.42]
Statistical Analysis 32: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2085, Mixed Models Analysis; Treatment Effect = -2.28, 80% CI 2-sided [-5.88 to 1.33]
Statistical Analysis 33: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 281; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6335, Mixed Models Analysis; Treatment Effect = 0.94, 80% CI 2-sided [-2.61 to 4.49]
Statistical Analysis 34: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1778, Mixed Models Analysis; Treatment Effect = -2.64, 80% CI 2-sided [-6.31 to 1.03]
Statistical Analysis 35: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.4027, Mixed Models Analysis; Treatment Effect = -0.70, 80% CI 2-sided [-4.33 to 2.94]
Statistical Analysis 36: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 309; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.7570, Mixed Models Analysis; Treatment Effect = 1.94, 80% CI 2-sided [-1.64 to 5.53]
Statistical Analysis 37: Comparison: CLG561 vs CLG561+LFG316; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1132, Mixed Models Analysis; Treatment Effect = -3.90, 80% CI 2-sided [-8.03 to 0.23]
Statistical Analysis 38: Comparison: CLG561 vs Sham Injection; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1965, Mixed Models Analysis; Treatment Effect = -2.71, 80% CI 2-sided [-6.80 to 1.37]
Statistical Analysis 39: Comparison: CLG561+LFG316 vs Sham Injection; Change from baseline at Day 337; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.6471, Mixed Models Analysis; Treatment Effect = 1.18, 80% CI 2-sided [-2.85 to 5.21]

9. Secondary Outcome: Average Change in BCVA From Baseline to the Period Day 281 to Day 337 as Measured by ETDRS
Description: BCVA was assessed using ETDRS testing at 4 meters. Day 281, Day 309, and Day 337 were averaged and compared to baseline. BCVA change was defined as a change in letters read from the baseline assessment. A positive change value indicates improvement. One eye (study eye) contributed to the analysis. No statistical analysis was conducted.
Time Frame: Baseline (Day 1), Day 281, Day 309, Day 337
Population: PPS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 30 | 35 | 34
letters | 3.0 (11.50) | 2.3 (13.25) | -0.3 (11.23)

10. Secondary Outcome: Average Change in LLVA From Baseline to the Period Day 281 to Day 337 as Measured by ETDRS
Description: LLVA was assessed at 4 meters using a neutral density filter to reduce chart luminance to 3 candelas/m2. Baseline is defined as the last measurement prior to first dose of treatment. Day 281, Day 309, and Day 337 were averaged and compared to baseline. BCVA change was defined as a change in letters read from the baseline assessment. A positive change value indicates improvement. One eye (study eye) contributed to the analysis. No statistical analysis was conducted.
Time Frame: Baseline (Day 1), Day 281, Day 309, Day 337
Population: PPS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 30 | 35 | 34
letters | 3.6 (11.04) | 0.4 (10.80) | -2.2 (17.01)

11. Secondary Outcome: Average LLVA Deficit (Letters) Change From Baseline at Day 281 to Day 337 as Measured by ETDRS
Description: LLVA was assessed at 4 meters using a neutral density filter to reduce chart luminance to 3 candelas/m2. A deficit in LLVA is defined as a loss in letters read from baseline. Baseline is defined as the last measurement prior to first dose of treatment. Day 281, Day 309, and Day 337 were averaged and compared to baseline. A negative change value indicates improvement (more letters read). One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 1), Day 281, Day 309, Day 337
Population: PPS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 30 | 35 | 34
letters | -0.6 (8.91) | 1.9 (12.96) | 1.9 (16.82)

12. Secondary Outcome: Percentage of Subjects With Letter Change in BCVA From Baseline up to Day 337 as Measured by ETDRS
Description: BCVA was assessed using ETDRS testing at 4 meters. Baseline is defined as the last measurement prior to first dose of treatment. BCVA change was defined as a change in letters read from the baseline assessment and is reported categorically. One eye (study eye) contributed to the analysis. No statistical analysis was conducted.
Time Frame: as for outcome 6
Population: FAS. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Number; unit: percentage of subjects
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
Number analyzed (Participants) | 35 | 37 | 38
percentage of subjects
  Change from BL at Day 2, ≥ 15 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 2, ≥ 15 letters | 2.9 | 2.8 | 0.0
  Change from BL at Day 2, ≥ 10 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 2, ≥ 10 letters | 8.6 | 5.6 | 2.7
  Change from BL at Day 2, ≥ 5 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 2, ≥ 5 letters | 20.0 | 27.8 | 10.8
  Change from BL at Day 2, ≤ -5 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 2, ≤ -5 letters | 20.0 | 5.6 | 18.9
  Change from BL at Day 2, ≤ -10 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 2, ≤ -10 letters | 5.7 | 2.8 | 5.4
  Change from BL at Day 2, ≤ -15 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 2, ≤ -15 letters | 5.7 | 0.0 | 5.4
  Change from BL at Day 8, ≥ 15 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 8, ≥ 15 letters | 2.9 | 5.6 | 0.0
  Change from BL at Day 8, ≥ 10 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 8, ≥ 10 letters | 23.5 | 5.6 | 5.3
  Change from BL at Day 8, ≥ 5 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 8, ≥ 5 letters | 29.4 | 27.8 | 21.1
  Change from BL at Day 8, ≤ -5 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 8, ≤ -5 letters | 8.8 | 8.3 | 13.2
  Change from BL at Day 8, ≤ -10 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 8, ≤ -10 letters | 5.9 | 5.6 | 5.3
  Change from BL at Day 8, ≤ -15 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 8, ≤ -15 letters | 0.0 | 2.8 | 0.0
  Change from BL at Day 15, ≥ 15 letters: number analyzed (Participants) | 33 | 36 | 38
  Change from BL at Day 15, ≥ 15 letters | 12.1 | 5.6 | 7.9
  Change from BL at Day 15, ≥ 10 letters: number analyzed (Participants) | 33 | 36 | 38
  Change from BL at Day 15, ≥ 10 letters | 18.2 | 11.1 | 15.8
  Change from BL at Day 15, ≥ 5 letters: number analyzed (Participants) | 33 | 36 | 38
  Change from BL at Day 15, ≥ 5 letters | 36.4 | 36.1 | 26.3
  Change from BL at Day 15, ≤ -5 letters: number analyzed (Participants) | 33 | 36 | 38
  Change from BL at Day 15, ≤ -5 letters | 6.1 | 8.3 | 15.8
  Change from BL at Day 15, ≤ -10 letters: number analyzed (Participants) | 33 | 36 | 38
  Change from BL at Day 15, ≤ -10 letters | 0.0 | 0.0 | 0.0
  Change from BL at Day 15, ≤ -15 letters: number analyzed (Participants) | 33 | 36 | 38
  Change from BL at Day 15, ≤ -15 letters | 0.0 | 0.0 | 0.0
  Change from BL at Day 29, ≥ 15 letters: number analyzed (Participants) | 34 | 37 | 38
  Change from BL at Day 29, ≥ 15 letters | 5.9 | 8.1 | 2.6
  Change from BL at Day 29, ≥ 10 letters: number analyzed (Participants) | 34 | 37 | 38
  Change from BL at Day 29, ≥ 10 letters | 20.6 | 18.9 | 10.5
  Change from BL at Day 29, ≥ 5 letters: number analyzed (Participants) | 34 | 37 | 38
  Change from BL at Day 29, ≥ 5 letters | 41.2 | 37.8 | 18.4
  Change from BL at Day 29, ≤ -5 letters: number analyzed (Participants) | 34 | 37 | 38
  Change from BL at Day 29, ≤ -5 letters | 11.8 | 5.4 | 13.2
  Change from BL at Day 29, ≤ -10 letters: number analyzed (Participants) | 34 | 37 | 38
  Change from BL at Day 29, ≤ -10 letters | 5.9 | 2.7 | 5.3
  Change from BL at Day 29, ≤ -15 letters: number analyzed (Participants) | 34 | 37 | 38
  Change from BL at Day 29, ≤ -15 letters | 0.0 | 0.0 | 2.6
  Change from BL at Day 30, ≥ 15 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 30, ≥ 15 letters | 12.1 | 5.6 | 8.1
  Change from BL at Day 30, ≥ 10 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 30, ≥ 10 letters | 18.2 | 13.9 | 13.5
  Change from BL at Day 30, ≥ 5 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 30, ≥ 5 letters | 45.5 | 33.3 | 24.3
  Change from BL at Day 30, ≤ -5 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 30, ≤ -5 letters | 6.1 | 11.1 | 13.5
  Change from BL at Day 30, ≤ -10 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 30, ≤ -10 letters | 0.0 | 2.8 | 5.4
  Change from BL at Day 30, ≤ -15 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 30, ≤ -15 letters | 0.0 | 2.8 | 2.7
  Change from BL at Day 57, ≥ 15 letters: number analyzed (Participants) | 35 | 37 | 37
  Change from BL at Day 57, ≥ 15 letters | 11.4 | 5.4 | 10.8
  Change from BL at Day 57, ≥ 10 letters: number analyzed (Participants) | 35 | 37 | 37
  Change from BL at Day 57, ≥ 10 letters | 22.9 | 16.2 | 16.2
  Change from BL at Day 57, ≥ 5 letters: number analyzed (Participants) | 35 | 37 | 37
  Change from BL at Day 57, ≥ 5 letters | 48.6 | 45.9 | 35.1
  Change from BL at Day 57, ≤ -5 letters: number analyzed (Participants) | 35 | 37 | 37
  Change from BL at Day 57, ≤ -5 letters | 8.6 | 13.5 | 13.5
  Change from BL at Day 57, ≤ -10 letters: number analyzed (Participants) | 35 | 37 | 37
  Change from BL at Day 57, ≤ -10 letters | 2.9 | 2.7 | 2.7
  Change from BL at Day 57, ≤ -15 letters: number analyzed (Participants) | 35 | 37 | 37
  Change from BL at Day 57, ≤ -15 letters | 0.00 | 0.00 | 0.00
  Change from BL at Day 85, ≥ 15 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 85, ≥ 15 letters | 8.6 | 5.6 | 8.1
  Change from BL at Day 85, ≥ 10 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 85, ≥ 10 letters | 28.6 | 13.9 | 13.5
  Change from BL at Day 85, ≥ 5 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 85, ≥ 5 letters | 45.7 | 38.9 | 24.3
  Change from BL at Day 85, ≤ -5 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 85, ≤ -5 letters | 8.6 | 16.7 | 13.5
  Change from BL at Day 85, ≤ -10 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 85, ≤ -10 letters | 0.0 | 5.6 | 2.7
  Change from BL at Day 85, ≤ -15 letters: number analyzed (Participants) | 35 | 36 | 37
  Change from BL at Day 85, ≤ -15 letters | 0.0 | 2.8 | 0.0
  Change from BL at Day 113, ≥ 15 letters: number analyzed (Participants) | 35 | 35 | 38
  Change from BL at Day 113, ≥ 15 letters | 8.6 | 2.9 | 7.9
  Change from BL at Day 113, ≥ 10 letters: number analyzed (Participants) | 35 | 35 | 38
  Change from BL at Day 113, ≥ 10 letters | 22.9 | 22.9 | 13.2
  Change from BL at Day 113, ≥ 5 letters: number analyzed (Participants) | 35 | 35 | 38
  Change from BL at Day 113, ≥ 5 letters | 40.0 | 40.0 | 23.7
  Change from BL at Day 113, ≤ -5 letters: number analyzed (Participants) | 35 | 35 | 38
  Change from BL at Day 113, ≤ -5 letters | 5.7 | 17.1 | 13.2
  Change from BL at Day 113, ≤ -10 letters: number analyzed (Participants) | 35 | 35 | 38
  Change from BL at Day 113, ≤ -10 letters | 2.9 | 8.6 | 5.3
  Change from BL at Day 113, ≤ -15 letters: number analyzed (Participants) | 35 | 35 | 38
  Change from BL at Day 113, ≤ -15 letters | 0.0 | 0.0 | 2.6
  Change from BL at Day 141, ≥ 15 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 141, ≥ 15 letters | 14.7 | 5.6 | 10.5
  Change from BL at Day 141, ≥ 10 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 141, ≥ 10 letters | 23.5 | 19.4 | 15.8
  Change from BL at Day 141, ≥ 5 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 141, ≥ 5 letters | 44.1 | 41.7 | 23.7
  Change from BL at Day 141 ≤ -5 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 141 ≤ -5 letters | 8.8 | 2.8 | 26.3
  Change from BL at Day 141, ≤ -10 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 141, ≤ -10 letters | 5.9 | 0.0 | 7.9
  Change from BL at Day 141, ≤ -15 letters: number analyzed (Participants) | 34 | 36 | 38
  Change from BL at Day 141, ≤ -15 letters | 2.9 | 0.0 | 0.0
  Change from BL at Day 169, ≥ 15 letters: number analyzed (Participants) | 32 | 37 | 37
  Change from BL at Day 169, ≥ 15 letters | 12.5 | 2.7 | 13.5
  Change from BL at Day 169, ≥ 10 letters: number analyzed (Participants) | 32 | 37 | 37
  Change from BL at Day 169, ≥ 10 letters | 21.9 | 13.5 | 18.9
  Change from BL at Day 169, ≥ 5 letters: number analyzed (Participants) | 32 | 37 | 37
  Change from BL at Day 169, ≥ 5 letters | 37.5 | 35.1 | 24.3
  Change from BL at Day 169, ≤ -5 letters: number analyzed (Participants) | 32 | 37 | 37
  Change from BL at Day 169, ≤ -5 letters | 21.9 | 18.9 | 10.8
  Change from BL at Day 169, ≤ -10 letters: number analyzed (Participants) | 32 | 37 | 37
  Change from BL at Day 169, ≤ -10 letters | 3.1 | 5.4 | 2.7
  Change from BL at Day 169, ≤ -15 letters: number analyzed (Participants) | 32 | 37 | 37
  Change from BL at Day 169, ≤ -15 letters | 0.0 | 2.7 | 0.0
  Change from BL at Day 197, ≥ 15 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 197, ≥ 15 letters | 15.2 | 2.8 | 10.8
  Change from BL at Day 197, ≥ 10 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 197, ≥ 10 letters | 30.3 | 13.9 | 18.9
  Change from BL at Day 197, ≥ 5 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 197, ≥ 5 letters | 45.5 | 41.7 | 32.4
  Change from BL at Day 197, ≤ -5 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 197, ≤ -5 letters | 21.2 | 19.4 | 16.2
  Change from BL at Day 197, ≤ -10 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 197, ≤ -10 letters | 9.1 | 11.1 | 10.8
  Change from BL at Day 197, ≤ -15 letters: number analyzed (Participants) | 33 | 36 | 37
  Change from BL at Day 197, ≤ -15 letters | 6.1 | 2.8 | 5.4
  Change from BL at Day 225, ≥ 15 letters: number analyzed (Participants) | 32 | 35 | 37
  Change from BL at Day 225, ≥ 15 letters | 21.9 | 8.6 | 8.1
  Change from BL at Day 225, ≥ 10 letters: number analyzed (Participants) | 32 | 35 | 37
  Change from BL at Day 225, ≥ 10 letters | 28.1 | 20.0 | 10.8
  Change from BL at Day 225, ≥ 5 letters: number analyzed (Participants) | 32 | 35 | 37
  Change from BL at Day 225, ≥ 5 letters | 37.5 | 45.7 | 21.6
  Change from BL at Day 225, ≤ -5 letters: number analyzed (Participants) | 32 | 35 | 37
  Change from BL at Day 225, ≤ -5 letters | 21.9 | 20.0 | 24.3
  Change from BL at Day 225, ≤ -10 letters: number analyzed (Participants) | 32 | 35 | 37
  Change from BL at Day 225, ≤ -10 letters | 9.4 | 5.7 | 16.2
  Change from BL at Day 225, ≤ -15 letters: number analyzed (Participants) | 32 | 35 | 37
  Change from BL at Day 225, ≤ -15 letters | 6.3 | 5.7 | 2.7
  Change from BL at Day 253, ≥ 15 letters: number analyzed (Participants) | 29 | 36 | 36
  Change from BL at Day 253, ≥ 15 letters | 17.2 | 5.6 | 13.9
  Change from BL at Day 253, ≥ 10 letters: number analyzed (Participants) | 29 | 36 | 36
  Change from BL at Day 253, ≥ 10 letters | 34.5 | 30.6 | 16.7
  Change from BL at Day 253, ≥ 5 letters: number analyzed (Participants) | 29 | 36 | 36
  Change from BL at Day 253, ≥ 5 letters | 44.8 | 38.9 | 16.7
  Change from BL at Day 253, ≤ -5 letters: number analyzed (Participants) | 29 | 36 | 36
  Change from BL at Day 253, ≤ -5 letters | 24.1 | 19.4 | 27.8
  Change from BL at Day 253, ≤ -10 letters: number analyzed (Participants) | 29 | 36 | 36
  Change from BL at Day 253, ≤ -10 letters | 3.4 | 13.9 | 19.4
  Change from BL at Day 253, ≤ -15 letters: number analyzed (Participants) | 29 | 36 | 36
  Change from BL at Day 253, ≤ -15 letters | 3.4 | 8.3 | 11.1
  Change from BL at Day 281, ≥ 15 letters: number analyzed (Participants) | 30 | 36 | 35
  Change from BL at Day 281, ≥ 15 letters | 23.3 | 8.3 | 8.6
  Change from BL at Day 281, ≥ 10 letters: number analyzed (Participants) | 30 | 36 | 35
  Change from BL at Day 281, ≥ 10 letters | 33.3 | 22.2 | 14.3
  Change from BL at Day 281, ≥ 5 letters: number analyzed (Participants) | 30 | 36 | 35
  Change from BL at Day 281, ≥ 5 letters | 43.3 | 44.4 | 28.6
  Change from BL at Day 281, ≤ -5 letters: number analyzed (Participants) | 30 | 36 | 35
  Change from BL at Day 281, ≤ -5 letters | 26.7 | 25.0 | 25.7
  Change from BL at Day 281, ≤ -10 letters: number analyzed (Participants) | 30 | 36 | 35
  Change from BL at Day 281, ≤ -10 letters | 6.7 | 22.2 | 20.0
  Change from BL at Day 281, ≤ -15 letters: number analyzed (Participants) | 30 | 36 | 35
  Change from BL at Day 281, ≤ -15 letters | 6.7 | 11.1 | 11.4
  Change from BL at Day 309, ≥ 15 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 309, ≥ 15 letters | 20.0 | 8.6 | 2.9
  Change from BL at Day 309, ≥ 10 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 309, ≥ 10 letters | 23.3 | 22.9 | 11.4
  Change from BL at Day 309, ≥ 5 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 309, ≥ 5 letters | 43.3 | 40.7 | 25.7
  Change from BL at Day 309, ≤ -5 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 309, ≤ -5 letters | 20.0 | 22.9 | 31.4
  Change from BL at Day 309, ≤ -10 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 309, ≤ -10 letters | 10.0 | 8.6 | 22.9
  Change from BL at Day 309, ≤ -15 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 309, ≤ -15 letters | 3.3 | 5.7 | 8.6
  Change from BL at Day 337, ≥ 15 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 337, ≥ 15 letters | 16.7 | 8.6 | 5.7
  Change from BL at Day 337, ≥ 10 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 337, ≥ 10 letters | 30.0 | 20.0 | 11.4
  Change from BL at Day 337, ≥ 5 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 337, ≥ 5 letters | 43.3 | 40.0 | 25.7
  Change from BL at Day 337, ≤ -5 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 337, ≤ -5 letters | 26.7 | 22.9 | 34.3
  Change from BL at Day 337, ≤ -10 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 337, ≤ -10 letters | 13.3 | 14.3 | 14.3
  Change from BL at Day 337, ≤ -15 letters: number analyzed (Participants) | 30 | 35 | 35
  Change from BL at Day 337, ≤ -15 letters | 6.7 | 11.4 | 5.7

13. Secondary Outcome: Total CLG561 Serum Concentrations up to Day 421
Description: Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method.
Time Frame: Baseline (Day 1), Day 2, Day 8, Day 15, Day 29, Day 85, Day 169, Day 253, Day 309, Day 337, Day 421
Population: PK Analysis Set. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CLG561 | CLG561+LFG316
Number analyzed (Participants) | 36 | 39
ng/mL
  Baseline: number analyzed (Participants) | 3 | 4
  Baseline | 0 (0) | 0 (0)
  Day 2: number analyzed (Participants) | 4 | 2
  Day 2 | 998 (471) | 475 (57)
  Day 8: number analyzed (Participants) | 5 | 3
  Day 8 | 821 (483) | 417 (90)
  Day 15: number analyzed (Participants) | 4 | 1
  Day 15 | 476 (76) | 428 (NA) — Standard deviation was not estimated due to low number of subjects with events.
  Day 29: number analyzed (Participants) | 2 | 1
  Day 29 | 181 (255) | 0 (NA) — Standard deviation was not estimated due to low number of subjects with events.
  Day 85: number analyzed (Participants) | 3 | 2
  Day 85 | 271 (236) | 0 (0)
  Day 169: number analyzed (Participants) | 9 | 10
  Day 169 | 294 (225) | 75 (160)
  Day 253: number analyzed (Participants) | 12 | 10
  Day 253 | 97 (178) | 36 (112)
  Day 309: number analyzed (Participants) | 14 | 13
  Day 309 | 161 (236) | 31 (113)
  Day 337: number analyzed (Participants) | 11 | 14
  Day 337 | 281 (242) | 54 (139)
  Day 421: number analyzed (Participants) | 17 | 18
  Day 421 | 0 (0) | 0 (0)

14. Secondary Outcome: Total LFG316 Serum Concentration up to Day 421
Description: as for outcome 13
Time Frame: Baseline (Day 1), Day 337, Day 421
Population: PK Analysis Set. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CLG561+LFG316
Number analyzed (Participants) | 39
ng/mL
  Baseline: number analyzed (Participants) | 1
  Baseline | 0 (NA) — Standard deviation was not estimated due to low number of subjects with events.
  Day 337: number analyzed (Participants) | 1
  Day 337 | 338 (NA) — Standard deviation was not estimated due to low number of subjects with events.
  Day 421: number analyzed (Participants) | 8
  Day 421 | 0 (0)

15. Secondary Outcome: Percentage of Subjects With Anti-CLG561 Antibodies up to Day 421
Description: Samples were collected and assessed for anti-CLG561 antibodies.
Time Frame: Baseline (Day 1), up to Day 421
Population: IG analysis set: All subjects in the safety analysis set with evaluable immunogenicity (IG) data and with no major protocol deviations that had an impact on the assessment of immunogenicity.
Measure: Number; unit: percentage of subjects
Arm/Group | CLG561 | CLG561+LFG316
Number analyzed (Participants) | 36 | 39
percentage of subjects | 0 | 7.7

16. Secondary Outcome: Percentage of Subjects With Anti-LFG316 Antibodies up to Day 421
Description: Samples were collected and assessed for anti-LFG316 antibodies.
Time Frame: Baseline (Day 1), up to Day 421
Population: as for outcome 15
Measure: Number; unit: percentage of subjects
Arm/Group | CLG561+LFG316
Number analyzed (Participants) | 39
percentage of subjects | 0

ADVERSE EVENTS:
Time Frame: Day 1 through study completion, an average of 336 days
Description: Adverse Events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Safety Analysis Set.
Groups:
- CLG561: All subjects exposed to CLG561 10 mg
- CLG561+LFG316: All subjects exposed to CLG561 5 mg + LFG316 5 mg
- Sham Injection: All subjects exposed to sham injection
Arm/Group | CLG561 | CLG561+LFG316 | Sham Injection
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/39 | 1/39
Serious Adverse Events (participants affected / at risk) | 5/36 | 5/39 | 7/39
Other Adverse Events (participants affected / at risk) | 27/36 | 31/39 | 29/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLG561 (N=36) | CLG561+LFG316 (N=39) | Sham Injection (N=39)
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Blindness (Eye disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLG561 (N=36) | CLG561+LFG316 (N=39) | Sham Injection (N=39)
Anterior chamber cell (Eye disorders) | 3 | 1 | 0
Anterior chamber flare (Eye disorders) | 2 | 0 | 0
Blepharitis (Eye disorders) | 1 | 3 | 5
Cataract nuclear (Eye disorders) | 0 | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 7 | 9 | 5
Conjunctival hyperaemia (Eye disorders) | 4 | 4 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 2
Dry age-related macular degeneration (Eye disorders) | 0 | 2 | 2
Dry eye (Eye disorders) | 3 | 0 | 2
Eye irritation (Eye disorders) | 2 | 2 | 4
Eye pain (Eye disorders) | 3 | 5 | 4
Iridocyclitis (Eye disorders) | 5 | 0 | 0
Metamorphopsia (Eye disorders) | 0 | 2 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 2
Photophobia (Eye disorders) | 0 | 2 | 0
Posterior capsule opacification (Eye disorders) | 1 | 2 | 1
Punctate keratitis (Eye disorders) | 2 | 2 | 0
Retinal haemorrhage (Eye disorders) | 3 | 4 | 1
Uveitis (Eye disorders) | 3 | 0 | 0
Visual acuity reduced (Eye disorders) | 12 | 8 | 5
Vitreal cells (Eye disorders) | 2 | 1 | 0
Vitreous detachment (Eye disorders) | 2 | 2 | 1
Vitreous floaters (Eye disorders) | 3 | 9 | 0
Vitreous opacities (Eye disorders) | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 3 | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 1 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3
Oral herpes (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1
Sinusitis (Infections and infestations) | 2 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Blood triglycerides increased (Investigations) | 0 | 0 | 2
Intraocular pressure increased (Investigations) | 4 | 4 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 3 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Renal cyst (Renal and urinary disorders) | 0 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 4 | 4 | 5
Hypotension (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT02515942/SAP_000.pdf
  • Study Protocol (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02515942/Prot_001.pdf